CLINICAL TRIAL: NCT00642005
Title: Humidification in Laparoscopic Colonic Surgery - A Double Blinded, Randomised Controlled Trial.
Brief Title: Humidification in Laparoscopic Colonic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Andrew G Hill, Professor of Surgery, University of Auckland, New Zealand
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Laphumid
Record Dates: First submitted 2008-03-17; First posted 2008-03-24 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Peritoneal Inflammation
Keywords: Humidification; Laparoscopy; Colon; Hemicolectomy; Warming
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Humidified and warmed carbon dioxide laparoscopic insufflation.
  Interventions: Procedure: Fisher and Paykel Humidifier (MR860)
- 2 (Placebo Comparator): Cold and dry carbon dioxide laparoscopic insufflation.
  Interventions: Procedure: Standard insufflation

INTERVENTIONS:
Procedure: Fisher and Paykel Humidifier (MR860) — Humidification to 98% relative humidity, and warming to 37 degrees C of laparoscopic insufflate. This will be done for the duration of the operation.
  Arms: 1
Procedure: Standard insufflation — No humidifier or warmer will be used (device switched off). This will deliver laparoscopic insufflate at 0% humidity and 20 degrees C.
  Arms: 2

SUMMARY:
Laparoscopic surgery allows surgeons to remove bowel via small incisions. To allow insertion of a camera and instruments, cold and dry gas is blown into the abdominal cavity. This project investigates the use of warmed, humidified gas in laparoscopic surgery. The hypothesis is that this will result in less damage to internal surfaces, and shorten recovery time. Previous studies have demonstrated positive outcomes in laparoscopic gallbladder operations. The investigators plan to study patients undergoing laparoscopic colon operations, as these operations are longer and the effect of humidification will be magnified. The investigators will enroll 74 patients: 37 will have the operation with cold dry gas, and 37 will have warm, humidified gas. The investigators will measure intraoperative heat loss, postoperative pain, fatigue, nausea and vomiting, and time to return of bowel function.

DETAILED DESCRIPTION:
The key determinants of a return to normal activity after major colorectal surgery are pain and fatigue. Our research group has an interest in enhancing perioperative care to reduce postoperative fatigue.

We have investigated the effect of peritoneal inflammation and the local production of cytokines on fatigue. Our data indicate that there is an association between the development of postoperative fatigue and the concentration of peritoneal cytokines following colorectal surgery. (Paddison, Hill - manuscript in submission). It is known that following surgery, there are two possible modes of communication between the cytokines and the brain. One is a hormonal routine by which the cytokines produced at the site of surgery enter the blood and proceed through cell surface receptors to act directly on the brain. The second method is a neural route represented by paracrine action of cytokines on primary afferent neurons that innervate the body site where the injury has taken place. In the abdominal cavity, the vagus nerve plays an important role in the latter form of communication. Vagal sensory neurons express large numbers of receptors for immune derived mediators, including a number of cytokines involved in inflammation and it has been shown that a major function of vagus may involve signaling immune and inflammatory situations. The vagus is unique as it has termination at the nucleus tractus solitarius (NTS) in the brain. The NTS is intensely activated following peripheral immune challenges and is also by far the most sensitive area in the brain following immune stimulation. The NTS projects monosynaptically to many regions of the brain which mediate sickness responses. Pro-inflammatory cytokines have been found in the blood, the skin, and the central nervous system after surgery and injury, however following major abdominal surgery such as colectomy these cytokines are found in very high concentrations in the peritoneal cavity. This local production of cytokines is far in excess of the amounts found in the serum suggesting an important local role and potentially a significant role in metabolic changes associated with colonic surgery. Therefore, inflammation and the consequent production of large concentrations of cytokines at the site of the surgery may activate the rich neurosensory vagal afferents to stimulate regions of the brain which mediate "sickness" responses. Therefore, it is feasible to hypothesize that strategies which lead to a reduction of the concentration of pro-inflammatory cytokines will lead to a reduction in post-operative fatigue.

In laparoscopic surgery, insufflated CO2 is delivered as defined by the United States Pharmacopoeia and National Formulary, which requires impurity of less than 200 parts per million, including water vapor. It is delivered at room temperature (21°C) with a relative humidity approaching 0%. Heat is lost by the body in warming and humidifying the cold, dry gas 1, and animal models have demonstrated that this can induce hypothermia. Initial human investigations showed that by simply heating the insufflating gas, core temperature was maintained and pain scores were improved. Additional findings showed heating and humidification helped to maintain core temperature in a porcine model 4. There is clinical evidence suggesting that heating and humidification can increase intraoperative core body temperature and reduce post-operative use of analgesia and pain scores for up to 14 days postoperatively. This intervention has also been linked significantly to an earlier return to normal activity in patients undergoing cholecystectomy.

Experimental studies have also shown that humidified gas is associated with less peritoneal and systemic inflammation compared to unhumidified gas. Furthermore, it has been demonstrated that use of warm, humidified gas is associated with a reduction in the concentration of peritoneal IL-6. The magnitude of this change is even larger than the effect seen after administration of anti-inflammatory agents in a similar setting. Significant reduction in other inflammatory peritoneal cytokines (TNF, IL-1) have also been observed in patients undergoing laparoscopic cholecystectomy with warmed CO2 insufflation gas.

Currently, there are no studies which have examined the effect of humidification in patients undergoing laparoscopic colonic surgery. We hypothesize that use of warm, humidified insufflation gas will lead to a reduction in hypothermia and concentration of peritoneal cytokines, with consequently decreased post-operative pain and fatigue, and earlier return to normal bowel function and activity. Our aim is to design and execute a double-blinded randomised controlled trial to test this hypothesis.

Research Design and Methods

Patients will be recruited from out-patient clinics across all three Auckland public hospitals. On the day of the operation, using opaque envelopes and computer generated random numbers; patients will be allocated into 2 groups. The intervention group will receive warm, humidified insufflation gas and control group will receive standard dry gas. Other intraoperative variables will be standardized and controlled. The patients, operating surgeons and other members of the clinical team will be blinded to the treatment given.

Using the data from a previous study measuring post-operative pain following colonic surgery; 37 patients are required in each group in to provide a 20% reduction in post-operative in hospital opiate use with alpha of 0.05 and power of 0.8. In order to achieve the required numbers we aim to enroll all patients undergoing laparoscopic colectomy from North Shore, Auckland and Middlemore Hospitals. Exclusion criteria:Patients under 15 years, acute cases, stoma formation (preop or intraop decision, decision to change to open surgery preoperatively (intraop conversions will be included as intention to treat), rectal lesions defined as less than 15cm from anal verge on imaging and/or sigmoidoscopy / colonoscopy, steroid dependence, inability to consent or answer SRS questions due to cognitive impairment or language barrier, ASA >= 4.

A reduction in postoperative morphine use forms the primary outcome of this study. Secondary outcomes include postoperative pain, fatigue, intraoperative heat loss and postoperative inflammatory response as measured by plasma and peritoneal pro-inflammatory cytokine concentration. Other outcomes that will be measured include nausea and vomiting, antiemetic use, and return of bowel function; with a reduction in these variables contributing to an endpoint of earlier return to normal activity.

Morphine equivalent analgesia usage will be documented in PACU, day of operation, day 1, day 2, and day 3. Visual analog scale measures of pain at rest will be obtained preoperatively, then at 2, 4, 8 and 12 hours, and days 1, 2, 3, 7, 14, 30, and 60 postoperatively.

Intraoperative temperature will be measured at 15min intervals using an naso-pharyngeal probe. A drain will be placed in the peritoneal cavity at the conclusion of surgery. On the morning following the operation, fluid from this drain as well as a simultaneous sample of blood will be collected, centrifuged and stored. Antioxidant levels will measures, and cytokine assays will be carried out by multiplexed cytometric bead immunoassays using the LINCOplex system (LINCO Research, St Charles, MO, USA). Drain fluid will be assayed for pro-inflammatory cytokines, IL-1a, TNF-a, IL-6, IL-8, IL-10 concentrations. Data will be acquired using a Luminex cytofluorimeter and analyzed using Luminex 100 IS software version 2.3 running a 4-parameter curve fit.

The SRS score will be used to measure surgical recovery, and will be administered preoperatively and also at days 1, 3, 7, 30, and 60. Anti-emetic use as well as time of return of normal bowel function (ability to eat and drink one complete hospital meal, passages of flatus or bowel motion and absence of nausea and vomiting) will also be recorded. Patients will be contacted on discharge to ascertain time to return of normal preoperative function.

ELIGIBILITY:
Inclusion Criteria:

* All patients 15 years and over undergoing elective laparoscopic colonic resection at all three auckland hospitals

Exclusion Criteria:

* Acute cases
* Stoma formation (preop or intraop decision)
* Decision to change to open surgery preoperatively (intraop conversions included as intention to treat)
* Rectal lesions defined as 15 cm from anal verge on imaging and/or sigmoidoscopy / colonoscopy
* Steroid dependence
* Inability to consent or answer SRS questions due to cognitive impairment or language barrier
* ASA >= 4

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Pain by visual analogue scale | preop, 2 hours, 4 hours, 8 hours, 12 hours, day 1, day 2, day 3, day 7, day 14, day 30, day 60
Morphine equivalent analgesia use | PACU, day of OT, day 1, day 2, day 3, total in hospital

SECONDARY OUTCOMES:
Intraoperative temperature by esophageal probe | 15 min intervals during surgery
Plasma and peritoneal cytokine concentration | Morning of surgery
Antiemetic use | PACU, day of OT, day 1, day 2, day 3
Return of bowel function - passage of flatus, bm, and eating first meal | daily
Any complications | Up to 3 months postoperatively
Surgical recovery by SRS | preop, day 1, day 2, day 3, day 7, day 30, day 60

OTHER OUTCOMES:
Small bowel obstruction | 5 year followup
  Admission to hospital within 5 years for small bowel obstruction, operative management or non-operative.
Survival | 5 year followup
  Overall survival and disease free survival at 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Hill, MBChB, MD, FRACS, Study Chair — University of Auckland, New Zealand
Locations (3):
- New Zealand (3):
  - Middlemore Hospital, Auckland, Otahuhu
  - Auckland City Hospital, Auckland
  - North Shore Hospital, Auckland

REFERENCES:
- [Derived] Sammour T, Hill AG. Five year follow-up of a randomized controlled trial on warming and humidification of insufflation gas in laparoscopic colonic surgery--impact on small bowel obstruction and oncologic outcomes. Int Surg. 2015 Apr;100(4):608-16. doi: 10.9738/INTSURG-D-14-00210.1. PMID 25875541